CLINICAL TRIAL: NCT06528002
Title: Hybrid Method Between Low-ratio Premixed Insulin and Short Acting Insulin in Fasting Type 2 Diabetic Patients in Ramadan: Safety and Efficacy
Brief Title: Hybrid Method Between Low-ratio Premixed Insulin and Short Acting Insulin in Fasting Type 2 Diabetic Patients in Ramadan
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Ahmed Mohamed, lecturer of internal medicine, Sohag University
Other Study IDs: Soh-Med-24-05--02PD.
Record Dates: First submitted 2024-07-15; First posted 2024-07-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-07

CONDITIONS: Continous Blood Glucose Monitoring; Calculation of Body Mass Index; Measurment of Blood Pressure
Keywords: type 2 DM.fasting in ramadan .insulin therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: type 2 diabetic patients take normal breakfast dose at Iftar and take 50% of dinner dose as short acting insulin at Suhoor with giving metformin dose after Suhoor even if giving once per day.
- Group 2: patients on regmin as recommendations of IDF take normal breakfast dose at Iftar and Reduce Suhoor dose by 20-50% of dinner premixed dose.

SUMMARY:
All healthy Muslim adults are required to observe the Ramadan fast, which is one of Islam's five pillars. People with Type 2 Diabetes Mellitus(T2DM). frequently fast throughout Ramadan. However, many Muslim patients insist on fasting in spite of medical warning. So, the investigators aim in the current study to assess safety and efficacy of our hybrid method using of low-ratio premixed insulin take at Iftar and short acting insulin take at Suhoor compare to last recommendation of IDF guideline of using low-ratio premix insulin regimens in type 2 diabetic patients who insist on Ramadan fasting.

DETAILED DESCRIPTION:
All healthy Muslim adults are required to observe the Ramadan fast, which is one of Islam's five pillars. People with Type 2 Diabetes Mellitus(T2DM). frequently fast throughout Ramadan.

Although fasting during Ramadan is said to have positive effects on diabetes patients, such as a reduction in excess body weight and an improvement in lipid profile, it can be linked to a slight increased risk for metabolic complications that need immediate attention, such as hypoglycemia and hyperglycemia, dehydration, and diabetic ketoacidosis (DKA)

Similarly, an increase in hyperglycemic episodes was also noted in another study conducted by the Benghazi Diabetes and Endocrine Centre (BDEC) on 493 T2DM patients fasting during Ramadan where 10.7% experienced hyperglycemia. Therefore, appropriate treatment adjustments including insulin regimen are necessary to avoid both hypo and hyperglycemia during Ramadan fasting.

T2DM patients well-controlled on premixed insulin or multiple doses injections should not fast, and they have the legitimate exemption for this. However, many Muslim patients insist on fasting inspite of medical warning. So, the investigators aim in the current study to assess safety and efficacy of our hybrid method using of low-ratio premixed insulin take at Iftar and short acting insulin take at Suhoor compare to last recommendation of IDF guideline of using low-ratio premix insulin regimens in type 2 diabetic patients who insist on Ramadan fasting.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian male and female Muslim patients,With T2DM, willing to fast Ramadan

  * . age ≥ 18 years old.
  * . type 2 diabetic patients treated with premixed insulin alone or combined with oral antidiabetic drugs (metformin, sulfonylurea: gliclazide, dipeptidyl peptidase 4 Inhibitor: sitagliptin or vildagliptin or thiazolidinediones/glitazones).

Exclusion Criteria:

* type 1 diabetic patients
* uncontrolled type 2 diabetics (HbA1c > 9; but they were included if insisting on fasting despite the detailed medical advice very high-risk diabetics (according to IDF 2021 classification)9
* newly diagnosed as diabetics (< 3 months)
* patients with previous ketoacidosis or hyperosmolar hyperglycemic states, recurrent or severe hypoglycemia within the past 2 months
* type 2 diabetic patients with hypoglycemic unawareness.
* Hospitalized patients, besides pregnant and lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will carry out on Muslim type 2 DM patients willing to fast Ramadan during the year 2024 attending outpatient clinic, Sohag faculty of medicine, Sohag university, Egypt.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
effect of hyprid method of insulin in type 2 diabetic patients during fasting in ramadan | 4 weeks after ramadan
  This is a study aiming to assess the safety and efficacy of our hybrid method compare to last recommendation of IDF guideline of using low-ratio premix insulin regimens in type 2 diabetic patients who insist on Ramadan fasting. and this done by measurement of blood glucose level 7 times daily to detect control of blood glucose during fasting in ramadan .then will measure fasting and postprandial blood glucose level after ramadan

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kasem Abdelal, lecturer, Study Chair — sohag university .faculty of medicine; Ahmed Faysal El_Rawy, lecturer, Study Chair — sohag university .faculty of medicine; Marwa zanaty Elsayed, lecturer, Study Chair — sohag university .faculty of medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided